CLINICAL TRIAL: NCT03152526
Title: A Randomized Trial Comparing CD3/CD19 Depleted or CD3 Depleted/CD56 Selected Haploidentical Donor Natural Killer (NK) Cell Based Therapy for Adults With Acute Myelogenous Leukemia Who Have Failed 1 or 2 Induction Attempts
Brief Title: CD3/CD19 Depleted or CD3 Depleted/CD56 Selected Haploidentical Donor Natural Killer (NK) Cell Based Therapy for AML Patients Not in CR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Miltenyi Biotec B.V. & Co. KG (Industry)
Collaborators: Masonic Cancer Center, University of Minnesota (Other); University of Chicago (Other); Ohio State University (Other)
Responsible Party: Sponsor
Organization: Miltenyi Biomedicine GmbH (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-2014-02; NCT03290664 (obsolete NCT alias)
Record Dates: First submitted 2017-02-28; First posted 2017-05-15 (Actual); Results first posted 2019-05-07 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-02

CONDITIONS: Acute Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Methods

STUDY DESIGN:
Intervention Model Description: In summary, the study will take place in two parts:
  Stage 1: Enroll 24 patients with 1:1 randomization for NK cell processing (CD3-/CD19- versus CD3-/CD56+) Stage 2: Enroll an additional 17 patients using the optimal NK cell product identified during stage 1.
  If neither product achieves success at the end of stage 1, the study will stop and the platform redesigned
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Single-arm trial (Other): Multi-center, open-label, single-arm, phase I/II clinical trial
  Interventions: Device: Interventions

INTERVENTIONS:
Device: Interventions — CliniMACS® CD3 and CD19 Reagent System
  Other Names: Devise

SUMMARY:
This is a phase II trial designed to test the safety and efficacy (complete response [CR]) of related donor HLA-haploidentical NK-cell based therapy for the treatment of acute myelogenous leukemia (AML).

Patients with newly diagnosed AML who failed to achieve a complete remission (CR) after one or two standard induction attempts receive after a preparative regimen of cyclophosphamide and fludarabine a single infusion of CD3-/CD19- NK cells or CD3-/CD56+ NK cells followed by a short course of Interleukin-2 (IL-2) to facilitate NK cell survival and expansion.

DETAILED DESCRIPTION:
This trial uses a Simon's two-stage design to estimate the complete remission rate at day +42 post NK cell infusion. The trial includes an initial randomized sub- study of 24 patients during stage 1 to choose which of the enriched NK cell products (CD3-/CD19- versus CD3-/CD56+) should be used to complete the trial based on successful in vivo NK cell expansion. This parameter is defined as 40% donor DNA and 40% of lymphocytes are NK cells at day 7 post infusion OR 20% donor DNA and 20% of lymphocytes are NK cells at day 14 post infusion. Twelve patients will be randomized to each product.

Enrollment Plan:

Stage 1: Enroll 24 patients with 1:1 randomization for NK cell processing (CD3-/CD19- versus CD3-/CD56+) Stage 2: Enroll an additional 17 patients using the optimal NK cell product identified during stage 1.

If neither product achieves success at the end of stage 1, the study will stop and the platform redesigned

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with acute myelogenous leukemia (except acute promyelocytic leukemia) and has failed one or two prior standard induction attempts. Failure is defined as:
* ≥ 30% bone marrow blasts with at least 20% cellularity at mid-cycle bone marrow biopsy or residual AML on subsequent~ day 28 bone marrow biopsy by morphology, flow, PCR or FISH
* Patients enrolling after only 1 failed induction attempt must meet at least one of the following additional eligibility criteria of high risk: ≥ 60 years of age adverse cytogenetics or molecular characteristics
* AML that progressed out of myelodysplastic syndrome (MDS) is eligible if the patient did not receive treatment directed at the MDS
* HLA-haploidentical related donor (aged 12 to 70 years)
* ≥ 18, but < 75 years of age
* Karnofsky performance status ≥ 60%
* Adequate organ function within 14 days of study registration (30 days for pulmonary and cardiac) as defined in section 4.5
* Ability to be off prednisone and other immunosuppressive drugs for at least 3 days prior to the NK cell infusion (excluding preparative regimen pre-meds)
* No prior hematopoietic transplant
* Not pregnant or lactating
* Sexually active females of childbearing potential and males with partners of child bearing potential must agree to use birth control

Exclusion Criteria:

* Pregnant or lactating as the treatments used in this study includes drugs that are FDA Pregnancy Category D.
* Acute leukemias of ambiguous lineage
* AML that transformed from previously treated myelodysplastic syndromes
* Prior hematopoietic transplant
* New or progressive pulmonary infiltrates on screening chest x-ray or chest CT scan that has not been cleared by Pulmonary. Infiltrates attributed to infection must be stable/improving (with associated clinical improvement) after 1 week of appropriate therapy (4 weeks for presumed or documented fungal infections)
* Uncontrolled bacterial, fungal, or viral infections including HIV - chronic asymptomatic viral hepatitis is allowed
* Known hypersensitivity to one or more of the study agents used

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-03-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Universtiy of Chicago, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CD3-/CD19- NK Cells Followed by IL-2: After a preparative regimen (day -6 to day -1) of fludarabine and cyclophosphamide participants receive allogeneic CD3-/CD19- NK Cell Product (NK Cell, CD3-/CD56+: ≥ 3-fold enrichment) on Day 0, followed by administration of interleukin-2 (after the NK cell infusion every other day for a total of 6 doses).
- CD3-/CD56+ NK Cells Followed by IL-2: After a preparative regimen (day -6 to day -1) of fludarabine and cyclophosphamide participants receive allogeneic CD3-/CD56+ Purified NK Cell Product (NK Cell, CD3-/CD56+: ≥ 70%) on Day 0, followed by administration of interleukin-2 (after the NK cell infusion every other day for a total of 6 doses).
Period: Overall Study
Arm/Group | CD3-/CD19- NK Cells Followed by IL-2 | CD3-/CD56+ NK Cells Followed by IL-2
Started | 0 (No participants were enrolled on this arm.) | 1 (One participant was enrolled on this arm.)
Completed | 0 (No participants were enrolled on this arm.) | 0 (The one participant enrolled on this arm withdrew from the study early.)
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: No participants were enrolled on the CD3-/CD19- NK cells arm. The study was closed due to poor enrollment.
Groups:
- Total: Total of all reporting groups
Arm/Group | CD3-/CD19- NK Cells Followed by IL-2 | CD3-/CD56+ NK Cells Followed by IL-2 | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Customized [Number; unit: years]
  Participant age (years) |  | 52 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 | 1
  Male |  | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint of the Study is Complete Remission (±3 Days)
Description: Both the number of patients with leukemia in complete remission and the number of patients with leukemia not in complete remission will be reported. Leukemia remission status will be assessed according to the Revised Recommendations of The International Working Group (J Clin Oncol 21:4642-4649, 2003).
Time Frame: On Day+42 (+/- 3 days) after NK cell infusion
Population: As a result of poor subject accrual (n=1), statistically relevant efficacy data cannot be defined according to the protocol.
Arm/Group | CD3-/CD19- NK Cells Followed by IL-2 | CD3-/CD56+ NK Cells Followed by IL-2
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: The Secondary Endpoint is the Expansion and Persistence of NK Cells to be Used for the Remainder of the Study.
Description: Successful expansion and persistence of NK cells is defined as ≥ 100 donor derived NK cells per µl blood.
Time Frame: Day+7 to Day+42 after NK cell infusion
Population: as for outcome 1
Arm/Group | CD3-/CD19- NK Cells Followed by IL-2 | CD3-/CD56+ NK Cells Followed by IL-2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: No participants were enrolled on the CD3-/CD19- NK Cells arm, therefore no participants on this arm were at risk of adverse events.
Arm/Group | CD3-/CD19- NK Cells Followed by IL-2 | CD3-/CD56+ NK Cells Followed by IL-2
All-Cause Mortality (participants affected / at risk) | 0/0 | 1/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/1
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CD3-/CD19- NK Cells Followed by IL-2 (N=0) | CD3-/CD56+ NK Cells Followed by IL-2 (N=1)
Serious adverse event (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Pulmonary edema, occurred prior to infusion of NK cell product and IL-2 and thus is not related to the IDE device or therapy; and is defined as a "serious adverse event" not related to IDE in Final Clinical Study Report without additional AE terms.
Serious adverse event (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Subject elected hospice care with disease progression and died of disease. The death was reported as a "serious adverse event" and stated as such on the Final Clinical Study Report without additional AE terms.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CD3-/CD19- NK Cells Followed by IL-2 (N=0) | CD3-/CD56+ NK Cells Followed by IL-2 (N=1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Chills, edema limbs, fever, injection site reaction (General disorders) | 0 | 1
Dyspnea, pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension, hypotension (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
As a result of poor subject accrual (n=1), statistically relevant efficacy data cannot be defined according to the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution conducted study as an independent contractor, supervised by the PI. PI may publish results provided that 12 months have elapsed since the completion of the study and sponsor has not initiated publication of a study report and at least 30 days prior to submission sponsor receives a draft to review. This study did not result in any publications.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-09): https://cdn.clinicaltrials.gov/large-docs/26/NCT03152526/Prot_SAP_000.pdf